CLINICAL TRIAL: NCT02163980
Title: Effect of Dexmedetomidine on the Characteristics of High Volume/Low Concentration Ropivacaine in a Caudal Block in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2011-0111
Record Dates: First submitted 2014-06-09; First posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Ambulatory Orchipexy
Keywords: dexmedetomidine; caudal block; children; children (1-6 years) undergoing ambulatory orchipexy
MeSH Terms: interventions — Saline Solution; Dexmedetomidine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caudal ropivacaine + normal saline (Placebo Comparator): 1.5ml kg-1 ropivacaine 0.15% with normal saline (Control group, n=40).
  Interventions: Drug: Caudal ropivacaine + normal saline
- Caudal ropivacaine + dexmedetomidine (Experimental): 1.5ml kg-1 ropivacaine 0.15% with dexmedetomidine 1 μg kg-1 (DEX group, n=40)
  Interventions: Drug: Caudal ropivacaine + dexmedetomidine

INTERVENTIONS:
Drug: Caudal ropivacaine + normal saline
  Arms: Caudal ropivacaine + normal saline
Drug: Caudal ropivacaine + dexmedetomidine
  Arms: Caudal ropivacaine + dexmedetomidine

SUMMARY:
The investigators perform this study to evaluate the effects of caudal Dexmedetomidine (DEX) added to high volume/low-concentration of ropivacaine in children undergoing orchiopexy.

ELIGIBILITY:
Inclusion Criteria:

* children undergoing ambulatory orchiopexy,
* ASA status I

Exclusion Criteria:

* mental retardation,
* developmental delay,
* neurological or psychiatric illness,
* coagulation disorder,
* spinal anomalies

Ages: 1 Year to 6 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2011-05; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
vital sign | up to 180 min after surgery
  systolic arterial pressure

SECONDARY OUTCOMES:
inhalation anesthetics requirements | up to 180 min after surgery
  end-tidal sevoflurane concentration required to maintain hemodynamic changes < 20% of the preoperative baseline

OTHER OUTCOMES:
incidence of agitation | up to 180 min after surgery
  number of patients
sedation score | up to 180 min after surgery
  three-point scale (0=eyes open spontaneously, 1=verbal stimulation, 2=physical stimulation
pain scores | up to 180 min after surgery
  Face Legs Activity Cry, Consolability scale (FLACC) Children's Hospital of Eastern Ontario Pain Scale (CHEOPS)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Univ. College of Medicine Dep. Of Anesthesiology, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Cho JE, Kim JY, Park SJ, Kil HK. The Effect of 1 microg/kg Dexmedetomidine Combined with High-Volume/Low-Concentration Caudal Ropivacaine in Children Undergoing Ambulatory Orchiopexy. Biol Pharm Bull. 2015;38(7):1020-5. doi: 10.1248/bpb.b15-00086. PMID 26133711